CLINICAL TRIAL: NCT07377305
Title: A Single-center, Prospective, Single-arm Clinical Study: Evaluation of the Efficacy and Safety of Transcranial Temporal Interference Stimulation (tTIS) for Neuropathic Pain in Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: Efficacy and Safety of Transcranial Temporal Interference Stimulation (tTIS) for Neuropathic Pain in Neuromyelitis Optica Spectrum Disorder (NMOSD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Jun Guo, MD, Associate Professor, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202512-50
Record Dates: First submitted 2026-01-08; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Current Stimulation (tTIS) Targeting Ventral Posterolateral Nucleus for Pain Treatment (Experimental): tTIS (10Hz envelope field, current intensity 2-4mA) targeted at ventral posterolateral nucleus (contralateral to the pain side) for 5 consecutive days (20 minutes/ day)
  Interventions: Device: 10Hz tTIS (2-4mA) Intervention

INTERVENTIONS:
Device: 10Hz tTIS (2-4mA) Intervention — tTIS (10Hz envelope field, current intensity 2-4mA)

SUMMARY:
This is an open-label, single-arm, single-center prospective pilot study to assess the efficacy and safety of transcranial temperol interference stimulation in patients with neuromyelitis optica spectrum disorder (NMOSD) complicated by neuropathic pain in China.

DETAILED DESCRIPTION:
Neuromyelitis optica spectrum disorder (NMOSD) is a rare but severe demyelinating condition that affects mainly adult patients. In the course of NMOSD, pain is a common accompanying symptom, aside from other symptoms such as visual impairment, limb weakness, limb numbness, and urinary and fecal dysfunction. Among these, neuropathic pain is the most common, affecting over 80% of patients with NMOSD. It occurs not only during the acute phase of NMOSD but also serves as the main form of chronic pain. Currently, there is no standard clinical protocol for the treatment of neuropathic pain, and the efficacy of analgesic drugs is limited. Transcranial temporal interference stimulation (tTIS) is emerging as a non-invasive therapeutic alternative to deep brain stimulation (DBS). Studies have shown that tTIS exerts a positive impact on neural function, including enhancing memory function and improving motor function. While it still remains underdeveloped about tTIS in the field of pain management. Based on this, we intend to conduct a small-sample prospective self-controlled study. By analyzing the baseline clinical characteristics, we will compare the changes in pain scale scores (Numerical Rating Scale [NRS], Visual Analog Scale [VAS]), Global Impression Scales, Short-Form McGill Pain Questionnaire, Painful Spasm Frequency Scale, and Hamilton Anxiety/Depression Scale scores before and after tTIS treatment. Through this, we aim to evaluate the efficacy and safety of this therapeutic approach in subjects suffered from NMOSD-related neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with NMOSD in accordance with the criteria of the International Panel for Neuromyelitis Optica Diagnosis (IPND).
* Patients were complicated with neuropathic pain, with a DN4 score ≥ 4.
* NRS score for pain ≥ 4 points, and neuropathic pain has persisted for more than 3 months.
* Patients receiving biological therapy and/or prednisone at a stable dose, with no adjustment of the treatment plan within 30 days before enrollment.
* Patients who have not adjusted any combination of standard analgesic drugs (including antiepileptic drugs, antidepressants, and opioid drugs) within 30 days before enrollment.
* Patients or their family members who have signed a written informed consent form.

Exclusion Criteria:

* Subjects participating in other clinical studies.
* Subjects who have used investigational drugs for pain control within 30 days before enrollment.
* Subjects with a concurrent diagnosis of peripheral neuropathy.
* Subjects with concurrent active central nervous system diseases.
* Subjects with cognitive or mental disorders.
* Subjects who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects with severe diseases related to the heart, liver, kidneys, or hematopoietic system.
* Subjects with implanted devices in the body (such as cardiac pacemakers, nerve stimulators, etc.).
* Subjects with a history of transcutaneous electrical nerve stimulation (TENS) allergy, latex allergy, or previous intolerance.
* Subjects with contraindications to MRI examination.
* Subjects with head skin lesions.
* Other medical conditions or situations that the researcher deems may affect the achievement of the study objectives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in numerical rating scale (NRS) score | Baseline, immediately after 5 consecutive treatments, 1 week after treatment, 2 weeks after treatment
  Patients are followed up and NRS score is determined. In general, the minimum and maximum scores of NRS are 0 and 10, respectively, with higher scores meaning a worse outcome.

SECONDARY OUTCOMES:
Change from baseline in visual analog scale (VAS) score | Baseline, immediately after 5 consecutive treatments, 1 week after treatment, 2 weeks after treatment
  Patients are followed up and VAS score is determined. In general, the minimum and maximum scores of VAS are 0 and 10, respectively, with higher scores meaning a worse outcome.
Change from baseline in patient global impression of change (PGIC) score | Immediately after 5 consecutive treatments, 1 week after treatment, 2 weeks after treatment
  Patients are followed up and PGIC score is determined. In general, the minimum and maximum scores of PGIC are 1 and 7, respectively, with higher scores meaning a worse outcome.
Change from baseline in short-form McGill pain questionnaire (SF-MPQ) score | Baseline, immediately after 5 consecutive treatments, 1 week after treatment, 2 weeks after treatment
  Patients are followed up and SF-MPQ score is determined. In general, the minimum and maximum scores of SF-MPQ are 0 and 45, respectively, with higher scores meaning a worse outcome.
Change from baseline in Penn spasm frequency scale (PSFS) score | Baseline, immediately after 5 consecutive treatments, 1 week after treatment, 2 weeks after treatment
  Patients are followed up and PSFS score is determined. In general, spasm frequency and spasm severity are evaluated. The minimum and maximum scores of spasm frequency are 0 and 4, respectively, with higher scores meaning a worse outcome. The minimum and maximum scores of spasm severity are 1 and 3, respectively, with higher scores meaning a worse outcome.
Change from baseline in Hamilton anxiety rating scale (HAMA) score | Baseline, immediately after 5 consecutive treatments, 1 week after treatment, 2 weeks after treatment
  Patients are followed up and HAMA score is determined. In general, the minimum and maximum scores of HAMA are 0 and 56, respectively, with higher scores meaning a worse outcome.
Change from baseline in Hamilton depression rating scale (HAMD) score | Baseline, immediately after 5 consecutive treatments, 1 week after treatment, 2 weeks after treatment
  Patients are followed up and HAMD score is determined. In general, the minimum and maximum scores of HAMD are 0 and 54, respectively, with higher scores meaning a worse outcome.
Adverse events | Baseline up to 2 weeks after treatment
  tTIS-related adverse events (AEs), such as headache, scalp irritation, rash, epilepsy, are evaluated and the rate of AEs is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China